CLINICAL TRIAL: NCT03904641
Title: Antimicrobial Photodynamic Therapy on Teeth With Molar Incisor Hypomineralization - a Randomized, Controlled, Clinical Trial
Brief Title: Antimicrobial Photodynamic Therapy on Teeth With Molar Incisor Hypomineralization
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HMIaPDT
Record Dates: First submitted 2019-04-04; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinical evaluations of complete removal of caries lesion, microbiological and radiographic analysis will be made by two blind examiners, who will not know to which group the participants belong.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aPDT + ART group (Experimental): In this group, both aPDT and ART will be performed.
  Interventions: Radiation: aPDT; Procedure: ART
- ART group (Experimental): In this group, only ART will be performed.
  Interventions: Procedure: ART

INTERVENTIONS:
Radiation: aPDT — For aPDT, PapacarieMblue (Fórmula e Ação) will be used. It will be left for 5 minutes in the cavity. The carious tissue will be removed and the application of the PapacarieMblue will be repeated. The tissue will then be irradiated in a single spot with a red laser, of wavelength of 660 nm, for 300 s, with the energy of 500mJ.
  Arms: aPDT + ART group
Procedure: ART — Removal of infected dentin with a curette only, followed by cavity cleaning and restoration with glass ionomer cement.

SUMMARY:
Molar Incisor Hypomineralization (MIH) is a change in the formation of dental enamel of systemic origin that affects at least one of the first four permanent molars and usually affects incisors. During the eruption, the affected surfaces tend to fracture, exposing the dentin, which causes excessive sensitivity in addition to making the region very susceptible to the appearance of carious lesions. The objective of this research will be to evaluate the clinical effect of antimicrobial photodynamic therapy (aPDT) in permanent teeth with severe and sensitive MIH. The methodology will be based on the selection of patients from 6 to 12 years of age with permanent molar teeth, randomly divided in two groups. The selected teeth should have MIH on the occlusal surface, indicated for clinical restorative treatment. In Group 1, aPDT will be applied for the treatment of infected dentin. Afterwards, the teeth will be restored with high viscosity glass ionomer cement. In Group 2, the removal of the softened dentin around the side walls of the cavity with sharp dentine curettes and posterior restoration with high viscosity glass ionomer cement will be carried out. All patients will have clinical and radiographic follow-up with a time interval of 6 and 12 months. The data obtained will be submitted to descriptive statistical analysis to evaluate the association of categorical variables. Chi-square test and Fisher's Exact test will be used, and to analyze the correlation between the continuous variables, Pearson correlation test will be applied. For the analysis of dentin density in the scanned radiographic images and the microbiological results for colony forming units, ANOVA and Kruskal-Wallis will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children, without systemic alterations;
* Collaborative children;
* Present at least one permanent molar with active and acute caries lesion in dentin, not exceeding 2/3 and involving only the occlusal, with direct vision and access, without clinical and radiographic signs and symptoms of pulp involvement.

Exclusion Criteria:

* Child with systemic impairment;
* Non-cooperative behavior;
* Carious lesion of Class II, III, IV or V type of Black;
* Clinically: carious lesion involving enamel, deficient restorations, small carious lesions in dentin (without access to hand excavators), occult caries lesions, clinical sign and/or symptom of pulp involvement, clinical impossibility of restoration;
* Radiographically: evidence of pulpal involvement, carious lesion extending beyond 2/3 of the dentin.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in dentin sensitivity | Baseline and immediately after treatment.
  Prior to removal of carious tissue, the volunteers will respond to the Visual Analogue Scale (VAS), following this protocol: gauze isolation of neighboring teeth and air jet in the tooth with MIH for 3 to 5 seconds. The evaluation of the sensitivity through the VAS will be repeated at the end of the procedure, after Atraumatic Restorative Treatment (ART).

SECONDARY OUTCOMES:
Change in colony forming units | Baseline and immediately after treatment.
  Microbiological specimens will be collected from the surface of the dentin before and immediately after the treatment, for later counting of colony forming units.
Change in dentin density | 6 and 12 months.
  The objective is to quantitatively determine the gray tones of the affected dentin region just below the glass ionomer restoration, whose radiographic control for visualization of the healthy dentin allows the clinical evaluator of the study to compare the treated groups with the density of the remaining dentin in discussion. The statistical analysis of the optical density will be made according to the mixed effects model.
Change in clinical aspect | 6 and 12 months.
  The retention of the material in the cavity and the presence of secondary caries will be evaluated.

REFERENCES:
- [Derived] Vieira LDS, Paschoal MAB, de Barros Motta P, Ferri EP, Ribeiro CDPV, Dos Santos-Pinto LAM, Motta LJ, Goncalves MLL, Horliana ACRT, Fernandes KPS, Ferrari RAM, Deana AM, Bussadori SK. Antimicrobial photodynamic therapy on teeth with molar incisor hypomineralization-controlled clinical trial. Medicine (Baltimore). 2019 Sep;98(39):e17355. doi: 10.1097/MD.0000000000017355. PMID 31574879